CLINICAL TRIAL: NCT06978543
Title: The Effect of a Device Developed for Flat or Inverted Nipples on Nipple Length, Breastfeeding and Feeding: A Randomized Controlled Study
Brief Title: The Effect of a Developed Device for Mother With Flat or Inverted Nipples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Zeynem YILDIRIM BALKAN, Assistant Professor and Principal Investigator, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TNKU-Z.BALKAN-3
Record Dates: First submitted 2025-04-21; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Inverted Nipple; Exclusive Breastfeeding
Keywords: Flat nipple; Inverted nipple; LATCH Score; Exclusive breastfeeding; Injector method
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The device developed for mothers with flat or inverted nipples who had just given birth, was compared with a control (injector method) group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Applications were made by the researcher (The intervention group:The device developed for mothers with flat or inverted nipples and the control group:injector method).
  Measurements (the diameter and length of the women's nipples, Baby's one time breastfeeding duration, Baby's one time attachment to the breast duration, LATCH scores, Babies exclusive breastfeeding duration in six months) were made by the nurse.
  The data were analysed by an independent statistician other than the researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DFIN Group (Experimental): The intervention group: A device developed for flat or inverted nipples (DFIN) was used. This device was developed by researchers. The developed device was printed on a 3D printer and applied to mothers. The way of using the tool is written in detail in the method.
  Interventions: Device: A Prototype Device Developed for Flat or Inverted Nipples (DFIN)
- Injector Group (Active Comparator): The syringe method used routinely in the unit was applied by the researcher to mothers immediately after delivery.
  Interventions: Device: Modified injector

INTERVENTIONS:
Device: A Prototype Device Developed for Flat or Inverted Nipples (DFIN) — This is a non-commercial, researchers-developed prototype breastfeeding aid (DFIN) designed for mothers with flat or inverted nipples. Produced using 3D printing, the device is made of biocompatible material and is not commercially registered. Prior to its application in patients, official approval for use was obtained from the Turkish Medicines and Medical Devices Agency (TITCK). DFIN was developed based on clinical experience and literature. Previous studies showed that warming the breast increases nipple temperature and enhances milk production. DFIN contains a 150-200 mL reservoir of warm water (39-41°C) to apply heat directly. It is anatomically designed to fit the breast and is kept in place for 10 minutes. Then the piston in the DFIN is pulled, with the mother's maximum comfort.
  Arms: DFIN Group
Device: Modified injector — The syringe method used routinely in the unit was applied by the researcher to mothers immediately after delivery. In this method, the thin part to which the needle is attached is cut with a sharp knife, the plunger is placed in this area and the syringe is applied to the flat or inverted nipple to create a vacuum
  Arms: Injector Group

SUMMARY:
Breast milk alone can meet all the elements necessary of babies during the first 6 months. However, some problems prevent breast milk from being taken, including concern about milk insufficiency, hyperlactation, clogged milk ducts, engorgement, mastitis, painful, injured/cracked nipples, flat or inverted nipples.

As there is insufficient nipple projection in mothers with flat or inverted nipples, it has been reported that babies have difficulty latching on to the breast and have problems breastfeeding. Also, it has been found that mothers with nipples shorter than 7 mm need more support. Many interventions are recommended to solve flat or inverted nipple problems.

In our study, a device developed for flat or inverted nipples was used by researchers. Thisa device developed for flat or inverted nipples was developed by researchers based on their experience and literature. This study was designed to evaluate the effects of the device developed for flat or inverted nipples for mother just already giving birth on nipple length, baby's attachment to the breast and breastfeeding duration, "LATCH Breastfeeding Assessment Tool" scores and and the duration of exclusive breastfeeding time in the first 6 months. The hypotheses of the study are as follows: (H1): Nipple length of mothers in the intervention gorup is longer. (H2): Babies in the intervention gorup would have a shorter attachment time on the breast. (H3): Babies in the intervention group have a longer duration of one breastfeeding. (H4): The LATCH breastfeeding diagnosis and evaluation score of the intervention group is higher. (H5): Babies in the intervention gorup have a longer exclusive breastfeeding time.

DETAILED DESCRIPTION:
This study employed a randomized controlled experimental design to evaluate the effectiveness of a device developed for flat or inverted nipples developed for mothers with flat or inverted nipples.

The study compared the effect of the flat or inverted nipple device with the injector method on nipple length, breastfeeding duration, exclusive breastfeeding duration and the LATCH Breastfeeding Diagnosis and Assessment Scale.

The research was conducted in an XXXXX University Hospital, Obstetrics and Gynecology Clinic. The population of the study consisted of 700 primiparous mothers who gave birth between November 2020 and November 2021. The inclusion criteria were that the mothers were aged 18 years or older, had normal or cesarean delivery at term, had a history of uncomplicated pregnancy or birth, and had a nipple length of 7 millimeter or less. Mothers with preterm and multiple births, babies with congenital anomalies, and women and babies with any health problems were excluded from the study.

The G*Power program was used to determine the required sample size. The power analysis used the results of a study in which a breastfeeding support program was implemented, evaluated with LACTH scores (experiment: 8.91±.98 and control: 7.78±1.3) and had an effect size of .98. In this study, it was aimed to create a change at the same effect level (.98 large effect) and it was calculated that there should be 29 mothers and babies per group (58 total) in the sample calculation made with 5% alpha margin of error (two-way) and and 90%. However, considering the possibility of loss during data collection, it was decided to include a total of 72 (36 per group) mothers and babies when it was calculated with 20% more for each group. During the follow-up, four mothers from both the interventio and injector groups were excluded for not participating in interviews, and one baby from the intervention group died. Thus, 31 the intervention gorup and 32 the injector group mothers and babies completed the study. Participants were randomly selected using the URN method, considered equivalent to full randomization. When a mother met the selection criteria, a random nurse assigned her to a group.

Research measurements

Information and follow-up form: This form included information such as mothers' age, education level, occupation, family income and type, pregnancy, and newborn's sex, birth weight and height, and Apgar Assessment score. The form was also used to record: nipple sizes, duration of time the baby was attachment to the breast and one breastfeeding. The nipple length of the mothers was measured. The researchers cut the ajutage off the 10 milliliter injectors and glued a millimetric transparent adhesive ruler on the cut. End then, the preperad injector placed on the nipple and the value seen on the transparent ruler was recorded as the nipple length. A paper ruler was used to measure the diameter of the nipples and aerolae of the mothers. The diameter of the nipple and areola was measured for each mother's a breast.

LATCH Breastfeeding Diagnosis and Assessment Scale form : The LATCH scale is a diagnostic tool developed based on the Apgar score assessment model. Each criterion of the LATCH Breastfeeding Diagnosis and Assessment Scale is scored 0, 1, 2. Breastfeeding success is assessed by adding up the scores. The highest score that can be obtained from the scale is 10 and the lowest score is 0. Increasing scores from the scale indicate breastfeeding success.

Nutrition form : This is the form that evaluates and records the baby's feeding types in terms of "Exclusive Breastfeeding, Breastmilk and Formula, Only Formula". This information is recorded at birth and the first, second, third, fourth, fifth, and sixth months. This is the form that evaluates and records the baby's feeding habits in terms of "breastmilk only, breastmilk and formula, and formula only".

In the study, the information and follow-up, the LATCH Scale and the nutrition form were performed by a lactation consultant nurse with 10 years of experience who was trained by the researchers.

Before the procedure: The purpose of the study was explained to the pregnant women who met the sample selection criteria by the researcher, and written consent was obtained from those who agreed to participate. After consent was obtained, participants were allocated to the intervention and injector groups in a randomized controlled manner. Demographic information of both groups was obtained. Immediately after delivery (Pre-application measurement), the diameter and length of the women's nipples, and the diameters of the areola were measured by a same clinical nurse and recorded on the information and follow-up form.

Application to the intervention group: The intervention group was used on the device immediately after giving birth. This device developed for flat or inverted nipples for mother. The use of the developed device is as follows: Firstly heated tap water (39-41 degrees Celsius) was added to the devices's water tank. Immediately after, the device was placed on the mother's breast and warm application was made with the device for 10 minutes. Meanwhile, the temperature of the breast and the water inside were measured at 2-3 minute intervals for 10 minutes. Before lifting the device from the breast, a vacuum was applied using the piston in the device at the maximum comfort of the mother. Then the device was removed from the breast. Right after the nipple was measured by the nurse. And the measurement was recorded on the "information and follow-up form (First post-application measurement)". Immediately after, the baby was placed on the mother's breast. Baby's one time breastfeeding and attachment to the breast duration were measured using a smartphone and recorded by the same nurse on the "information and follow-up form (First post-application measurement)". At the same time, breastfeeding success was evaluated using the LATCH Breastfeeding Diagnosis and Assessment Scale by observing the mother and baby by the same nurse (First post-application measurement). The hospital's routine practice is to breastfeed each baby every 2 hours after birth. Therefore, the second and third application and measurement with the device were made in the same way just before the next breastfeeding of the mother in the group (second and third post-application measurements).

Application to the injector group: The syringe method used routinely in the unit was applied by the researcher to mothers immediately after delivery. In this method, the thin part to which the needle is attached is cut with a sharp knife, the plunger is placed in this area and the syringe is applied to the flat or inverted nipple to create a vacuum. The syringe method was also used the same way in this study. After removing the injector from the breast, the nipple was measured the nurse. The measurement was recorded on the "information and follow-up form (first post-application measurement)" by the same nurse. Immediately after, the baby was placed on the mother's breast. Baby's one time breastfeeding and attachment to the breast duration were measured using a smartphone and recorded by the same nurse on the "information and follow-up form (first post-application measurement)". At the same time, breastfeeding success was evaluated using the he LATCH Breastfeeding Diagnosis and Assessment Scale by observing the mother and baby by the same nurse (first post-application measurement). The hospital's routine practice is to breastfeed each baby every 2 hours after birth. Therefore, the second and third application and measurement with the injector method were made in the same way just before the next breastfeeding of the mother in the group (2nd and 3rd post-application measurements).

Mothers and babies in both groups were contacted by the same nurse at 1, 2, 3, 4, 5 and 6 months after discharge and asked whether the babies had been exclusively breastfed. The information obtained was recorded on the Nutrition form.

ELIGIBILITY:
Inclusion Criteria:

The mothers:

* were aged 18 years or older,
* had normal or cesarean delivery at term,
* had a history of uncomplicated pregnancy or birth,
* had a nipple length of 7 mm or less.

Exclusion Criteria:

The mothers:

* Mothers with preterm and multiple births,
* babies with congenital anomalies,
* women and babies with any health problems were excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
The mean nipple lengths of the mothers | Through study completion, an average of 1 year
  Immediately after the interventions on the mother's nipples, the nipple length was measured by the nurse.
The LATCH score | Through study completion, an average of 1 year
  Immediately after the interventions on the mother's nipples, the LATCH score was measured by the nurse. LATCH Breastfeeding Diagnosis and Assessment Scale form : The LATCH scale is a diagnostic tool developed based on the Apgar score assessment model. Each criterion of the LATCH Breastfeeding Diagnosis and Assessment Scale is scored 0, 1, 2. Breastfeeding success is assessed by adding up the scores. The highest score that can be obtained from the scale is 10 and the lowest score is 0. Increasing scores from the scale indicate breastfeeding success.
The duration of baby's attachment to the breast | Through study completion, an average of 1 year
  Immediately after the interventions on the mother's nipples, the duration of baby's attachment to the breast was measured by the nurse.
The duration of baby's one time breastfeeding | Through study completion, an average of 1 year
  Immediately after the interventions on the The duration of baby's one time breastfeeding was measured by the nurse.
Feeding Taypes of Babies | Through study completion, an average of 1 year.
  Mothers and babies in both groups were contacted by the same nurse after discharge and asked whether the babies had been exclusively breastfed.

CONTACTS AND LOCATIONS:
Overall Officials: Serap BALCI, PhD,Prof., Principal Investigator — ISTANBUL UNİVERSİTY CERRAHPAŞA
Locations (1):
- Tekirdag Namık Kemal University, Tekirdağ, Suleymanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The full plan and results of the research can be seen when the article is published.